CLINICAL TRIAL: NCT06628271
Title: Breath-holding Spells and Its Management: a Prospective Study on Patient and Disease Characteristics, Evaluation of Novel Guidelines, Parental Handling, and Long-term Follow-up in Breath-holding Spells
Brief Title: Breath-holding Spells and Its Management Study
Acronym: BAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-03363-01
Record Dates: First submitted 2024-09-16; First posted 2024-10-04 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Breath-holding Spell
Keywords: disease definition; electrocardiography; iron deficiency anemia; long QT syndrome; parental support
MeSH Terms: conditions — Anemia, Iron-Deficiency; Long QT Syndrome

STUDY DESIGN:
Intervention Model Description: Inclusion upon suspicion of Breath Holding Spell. Thereafter, allocation to either the group that has a defined typical Breath Holding spell, or the alternative (parallel) group that is not diagnosed with a typical Breath Holding Spell. Subsequent management of study subject in the Typical Breath Holding Spell group according to the management algorithm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Typical spells (Other): Patients with typical spells should be investigated according to our guidelines
  Interventions: Diagnostic Test: Guidelines
- Non-typical spells (No Intervention): Patients with non-typical spells will be investigated individually, as it is done today

INTERVENTIONS:
Diagnostic Test: Guidelines — Participant with typical spells will be investigated according to our guidelines. These include that participants with heredity for or signs and symptoms of cardiac disease will be subjected to an ECG and participants with two or more spells should be subjected to blood tests for anemia and iron deficiency
  Arms: Typical spells

SUMMARY:
The goal of this prospective population-based study is to evaluate the new disease description and management guidelines for breath-holding spells in children (Hellström Schmidt et al, Acta Paediatrica 2024) below the age of 5 years in southern Sweden. The main questions it aims to answer are:

* Does the disease description and management guidelines lead to the expected reduction in diagnostic interventions and are the clinical managements guidelines safe to use?
* If iron supplementation is given, does it reduce the frequency and severity of the spells?
* What information and support does parents to children with breath-holding spells need?

Participants will undergo evaluation by a medical doctor and if typical breath-holding spells are diagnosed, be managed according to the new guidelines. If iron deficiency is found, iron supplementation is recommended. Digital surveys will be distributed and parents of patients with frequent spells will be eligible for participation in an interview sub-study.

DETAILED DESCRIPTION:
Please see the Study plan among the documents.

ELIGIBILITY:
Inclusion Criteria:

* Below 5 years of age
* resident in Region Skåne (Sweden)
* suspected breath-holding spell

Exclusion Criteria:

* previous investigation for breath-holding spell (previous spells are not a reason for exclusion)

Ages: 0 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Safety of the guidelines | From date of inclusion to end of follow up at 36 months
  The number of wrongful and missed diagnoses (definition: managed and diagnosed as breath-holding spells at physician assessment within study but later found to be another cause for the symptoms, like long QT syndrome or epilepsy).
Usability of the guidelines | From date of inclusion until last diagnostic intervention, expected to be within 2 weeks from inclusion.
  Assessed according to the following:
  * Number of patients with a diagnostic interventions for each intervention in the guidelines: ECGs and bloodtests.
  * Number of found pathologies for each intervention (blood tests and ECGs) - for patients with typical spells handled according to the guidelines and those with non-typical spells managed individually. This includes a retrospective assessment of ECG (a complete assessment including rythm, long QT syndrome, AV-block, ST-segment changes) and blood test results (for anemia and iron deficiency; i.e. values outside of the age adapted normal range).
  * Retrospective analysis of the clinical doctors compliance with managment guidelines, evaluated through the number of interventions for each patient that were not recommended in the guidlines (for instance number of EEGs).
Usability of the disease definition | From the inclusion date until end of physicians assessment
  Assessed according to the following:
  * Adherence to the the prespecified definition of typical spells through comparison of clinical physicians assessment and a retrospective assessment by study physician, i.e. the number of cases with a discrepant judgment of the clinical presentation.
  * The number of typical spells compared to the number of non-typical spells and other diagnsoses.
  * Compilation of patient and spell characteristics (defined in the variable list in the attached documents) and comparison with the current definition of typical spells.

SECONDARY OUTCOMES:
Need of information and support to parents | From 6 months after inclusion until interview is performed (expected to be within three months of six month digital survey)
  Through interview study (qualitative study) gather information on given information and support and their need for more information and support. Will be conducted on parents of children with more than 5 spells in total at the 6 month follow up (assessed as frequent spells).
Effect of iron supplement treatment on spell frequency and severity | From the date of inclusion until evaluation of iron treatment, most probably within 12 months from inclusion.
  In cases of iron treatment (initiated by the clinical physician). Assessed according to the following:
  * Comparison of spell frequency (number of spells/time unit) before start of treatment, during treatment and after completion of treament.
  * Comparison of spell severity (simple or severe spells defined as spells without and with loss of consciousness) before start of treatment, during treatment and after completion of treament.
  * Anemia and iron deficiency blood test values (Hb, MCV, reticulocytes, ferritin, CRP if signs of infection, iron, iron saturation and transferrin) comparison between patients with effect of iron treatment on spell frequency and severity, versus the group without a clinical effect of iron treatment.
  * Patient compliance for iron supplementation as per survey question with answer altneratives yes/no/don't know

OTHER OUTCOMES:
Natural course of the spells through long term follow-up | 36 months
  Assessed according to the following parameters, through digital surveys:
  * Spells during the last 3 months (yes or no)
  * Number of spells the previous month (0, 1, 2-5, 6-10, >10)
  * Total number of spells (free text)
  * Uncontactable or unconscious (=severity of spells) (Yes, No, Don't know)
  * Alterations in spell semiology? (Yes, No, Don't know)
Contact with health care during long term follow-up | 36 months
  Evaluation of the following questions:
  1. Do parents follow the advice to reach out to health care if the spell semiology change?
  2. Planned follow up?
  Above questions are assessed in a digital survey:
  - Further contact with healthcare. Answer alternatives: (Yes, No, Don't know). If yes: (acute or planned)
Burden of care | 36 months
  Will be assessed through a combined evaluation of the following variables:
  * Number of acute health care visits
  * Number of planned health care visits including follow-up appointments over phone
  * Number of over-night hospital stays (number of nights)
  * Number of ambulance rides to the hospital
Dietary impact on iron status | From inclusion to blood test results, within 2 weeks from initial visit
  At first visit, parents will answer questions on the child and family's diet in a questionnaire, to evaluate a possible association between diet and iron status (and further, to breath-holding spell frequency and severity).
  The questions are as follows:
  * Mark all alternatives that is correct about your childs diet: (breatmilk/formula/cow's milk/taste portions/family meals)
  * Does your child drink more than 3 dl of cow's milk per day? (yes/no)
    > If yes, estimate the amount of cow's milk your child drink during a day in dl: (a number in free text)
  * Do you eat vegetarian or vegan food only? (yes/no)

CONTACTS AND LOCATIONS:
Locations (12):
- Sweden (12):
  - Barn- och ungdomsmedicinmottagning Eslöv, Eslöv
  - Capio Barnavårdscentral Kristianstad, Kristianstad
  - Barnläkargruppen Sparta, Lund
  - Skåne University Hospital, Lund
  - Barnläkargruppen Sparta, Malmo
  - BVC Bambino Hyllie, Malmo
  - BVC Bambino Lindängen, Malmo
  - BVC Bambino Mobilia, Malmo
  - Skåne University Hospital, Malmo
  - Barn- och ungdomsmedicinmottagning Simrishamn, Capio närsjukhus, Simrishamn
  - Familjecentralen Björken, BVC Sjöbo, Sjöbo
  - Lasarettet i Ystad, Ystad

IPD SHARING:
Plan to Share IPD: Undecided
Data will be share as far as the Swedish law (concerning patient confidentiality) and ethical considerations allows. Decisions will be made from case to case depending on what data are inquired for.

REFERENCES:
- [Background] Hellstrom Schmidt S, Smedenmark J, Jeremiasen I, Sigurdsson B, Eklund EA, Pronk CJ. Overuse of EEG and ECG in children with breath-holding spells and its implication for the management of the spells. Acta Paediatr. 2024 Feb;113(2):317-326. doi: 10.1111/apa.17020. Epub 2023 Oct 31. PMID 37905418
- [Background] Hellstrom Schmidt S, Tedgard U, Pronk CJ. Breath-holding spells occur disproportionately more often in children with transient erythroblastopenia. Acta Paediatr. 2016 Sep;105(9):1088-93. doi: 10.1111/apa.13428. Epub 2016 Apr 29. PMID 27060698

DOCUMENTS (2):
  • Study Protocol (2024-10-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT06628271/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-16): https://cdn.clinicaltrials.gov/large-docs/71/NCT06628271/SAP_001.pdf